CLINICAL TRIAL: NCT04957251
Title: Does the Anterior or Posterior Approach to the Hip Provide Superior Functional Recovery After Recovery After Performing Hip Hemiarthroplasty
Brief Title: Anterior vs Posterior Approach for Hip Hemiarthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 150819-1
Record Dates: First submitted 2018-03-23; First posted 2021-07-12 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anterior approach (Experimental): Patient's undergoing an anterior approach to the hip
  Interventions: Procedure: anterior approach to the hip
- Posterior Approach (Active Comparator): Patient's undergoing an posterior approach to the hip
  Interventions: Procedure: posterior approach to the hip

INTERVENTIONS:
Procedure: anterior approach to the hip — anterior hip hemiarthroplasty
  Arms: Anterior approach
Procedure: posterior approach to the hip — posterior hip hemiarthroplasty
  Arms: Posterior Approach

SUMMARY:
Randomized trial to evaluate the role of the anterior vs posterior approach regarding hemiarthroplasty of the hip. The Investigators' hypothesis is that the muscle sparing anterior approach may result in improved function in the short term, which may allow shorter hospital stay and quicker return to prior level of function.

DETAILED DESCRIPTION:
Background

In patients who sustain a displaced femoral neck fracture, who do not meet criteria for total hip arthroplasty, the recommendations are made for a hemi-arthroplasty of the hip. There are multiple surgical approaches that can be used including the anterior approach to the hip and the posterior approach to the hip. The most widely performed approach to the hip when performing a total hip arthroplasty or hemi-arthroplasty has been the posterior approach. However, multiple approaches exist including posterior approach, direct lateral approach, anterolateral approach and direct anterior approach. There is not a consensus about which approach is the most appropriate or best for patients. The decision for approach is widely decided by the surgeon and is based on experience and preference of the surgeon. Recent advances in the anterior approach to the hip have found improved results with regards to functional status and decreased complications when compared to the posterior approach for total hip arthroplasty. There have been several retrospective studies comparing the anterior vs. posterior approach for hemi-arthroplasty with regards to treatment of femoral neck fractures. These studies have shown conflicting results with regards to which approach is superior. Retrospective studies have shown decreased dislocation rate with the anterior approach, but increased operative time and increased rate of infection with anterior approach as well. To date, there have been two prospective studies performed comparing the anterior and posterior approach for hemi-arthroplasty, one in Japan and one in France, both of which showed decreased dislocation rates but did not display long term functional improvement comparing the two approaches. Both of these studies' patient population and protocol differ greatly from standard of care in the United States. To date, there have been no prospective randomized controlled trials evaluating the functional advantage of the anterior vs. the posterior approach when performing hip hemi-arthroplasty procedure for femoral neck fractures in the United States. It is our hypothesis that the anterior approach will provide superior functional results as a product of the decreased damage to soft tissue and restoration of normal anatomy.

Objectives:

There are several objectives of this study.

The main objective of this study is to evaluate the functional status of each patient using a Harris Hip Score to evaluate both function and pain comparing the anterior vs. the posterior approach for hemi-arthroplasty at 6 months.

Secondary objectives of this study include:

* time to ambulation post operatively
* rate of complications including infection, nerve palsy, and DVT/PE
* operative time
* rate of dislocation
* periprosthetic fracture
* mortality
* return to preoperative mobility status
* blood loss

Significance:

The results of this study would either confirm the retrospective data that currently exists showing no difference in functional outcomes between the two approaches or demonstrate a superior functional status with either the anterior or posterior approach for hip hemi-arthroplasty. Of which, logically and anecdotally, the Investigators' believe will be the anterior approach. With this research, theInvestigators' believe the anterior approach can become the standard of care for the surgical technique with regards to hemi-arthroplasty for hip fractures

Eligible patients:

Eligible patients will include all patients that were previously ambulatory at some level who sustain a displaced femoral neck fracture that given functional status, age, and comorbidities will require a hemi-arthroplasty for definitive treatment. Ages 65-99

Patients who will be excluded from the study are all patients who are non ambulatory at baseline.

Design:

Patients who meet eligibility criteria will be offered to participate in the study. Once the patient consents, the participants will be randomized to receive either the anterior or posterior approach for hemi-arthroplasty of the hip. After surgery, the participant will undergo standard postoperative care (hip precautions) with data collected from the electronic health record and from standard hospital care including rounding. The participant will then follow up at appropriate standard interval with the main endpoint of 6 months where Harris Hip Scores will be used to judge the participant's functional status as well as pain relief.

Analysis of the collected data will occur at intervals of 50 patients to evaluate trends or statistical significance.

Monitoring Participants:

If at any time during this study the participant or medical decision maker decides to no longer participate in the study, the participant will be removed from the study and will continue to undergo standard treatment for their condition.

Consent:

Consent will be obtained so long as the participant meets the appropriate criteria listed above and will be given a detailed informed consent document outlining the purpose of the study and associated risks and benefits.

Human Subject Protections:

There is currently no widely accepted technique based on outcomes with regards to operative approach for hip hemi-arthroplasty, nor is there a standard approach for total hip arthroplasty. Therefore, the participant will not have to do anything different from an intervention standpoint and therefore are not at any increased risk based on our study protocol. All participants will receive treatment of hip fracture in an appropriate fashion. They will be asked standard postoperative questions during their stay and will undergo standard follow up. The only change from current standard of care in follow up will include the primary investigator performing a Harris Hip questionnaire and assessment at each postoperative visit.

With regards to selection, the only criteria will be a baseline ambulatory status prior to sustaining a displaced femoral neck fracture. The participants who are demented will be included in the study because a large percentage of patients who sustain femoral neck fractures and require a hemi-arthroplasty have some baseline dementia. These participants will only be included if a medical power of attorney or appropriate medical decision maker is available.

Analysis

Data will be collected and analyzed after 50 participants using a student t-test analysis to evaluate for statistical significance or tends. The goal of 200 patients is to obtain the largest prospective controlled trial to date. Analysis every 50 is based off of previous literature that showed statistical significance near 50 patients in some categories including dislocation.

Adverse Events Reporting

This study is a single surgeon study that is not blinded and all adverse events outside of the expected complications associated with hip hemi-arthroplasty will be reported immediately to the IRB board.

Patient confidentiality

The only PHI data that will be kept will be the FIN number to pull information from the electronic health record during analysis. This is necessary as a means to be able to accurately report lab values, operative times, and other pertinent information from their hospital stay. Otherwise, all hard copy data will be locked in a safe location, and all electronic data will be password protected.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will include all patients that were previously ambulatory at some level who sustain a displaced femoral neck fracture that given functional status, age, and comorbidities will require a hemi-arthroplasty for definitive treatment.
* Ages 65-99

Exclusion Criteria:

* Patients who will be excluded from the study are all patients who are non ambulatory at baseline.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes | 1 year
  Harris Hip Score. Score ranges from 0-100 The higher the HHS, the less dysfunction. A total score of <70 is considered a poor result; 70-80 is considered fair, 80-90 is good, and 90-100 is an excellent result

IPD SHARING:
Plan to Share IPD: Yes
Database that is kept on site that may be reviewed.